CLINICAL TRIAL: NCT00792402
Title: Implementation Process and Impact of the Heart Failure Electronic Clinical Guideline in the Catalan Health Institute Primary Care Health Board
Brief Title: Computerized Guideline in Heart Failure: Implementation Process and Impact Evaluation
Status: Completed | Type: Observational
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Catalan Institute of Health (Other Government)
Responsible Party: Sponsor
Other Study IDs: PI07/91020
Record Dates: First submitted 2008-11-17; First posted 2008-11-18 (Estimated); Last update posted 2011-11-23 (Estimated); Status verified 2011-11

CONDITIONS: Chronic Heart Failure
Keywords: chronic heart failure; Computerized clinical guidelines; Primary care

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1 control group: Computerized data collection of outcome measures in usual care
- 2 intervention group: Computerized data collection of outcome measures and interviews to clinicians which are using a computerized Heart Failure guideline in their daily practice.

SUMMARY:
Objective: To assess the effectiveness of implementation process of an electronic Heart Failure guideline in primary care in the city of Barcelona.

DETAILED DESCRIPTION:
Design: Two types of design will be applied, according to the specific aims. On the one hand it is a cross-sectional and a qualitative study, on the other hand it is quasi-experimental study. Pre-post intervention with a control group, as well as, of repeated measures in the intervention group

ELIGIBILITY:
Inclusion Criteria:

* general and nurse primary care practitioners working in Barcelona and Girona for the Health Catalan Institute.
* Managers involved in implementation process for the computerised clinical guideline in Barcelona from the Health Catalan Institute.
* patients with diagnoses of Heart Failure according to ICD-10 according to general practice clinical records.

Exclusion Criteria:

* Managers and general and nurse primary care practitioners working in Barcelona health Centres where there were any other quality improvement project related to Heart failure at the time of the intervention which we are evaluating. Managers from the control group (Girona).
* patients with a mental health disorder or terminal illness

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Setting: 20 general practices in Barcelona (intervention group),with an assigned population of 558515 inhabitants and Girona (control Group) with 23 general practices, and an assigned population of 480827.In 2007, the intervention region had a rate of 1499 patients per GP and from 16 to 52 thousand listed patients per practice with and average of attending rate of 68%, and the control region had a rate of 1558 patients per GP and from 4 to 47 thousand listed patients per practice with and average of attending rate of 76%.
  Subjects: Managers and general and nurse practitioners from Barcelona and Girona primary care practices included in the study. Patients with diagnoses related to Heart Failure.
Sampling Method: Non-Probability Sample
Enrollment: 13008 (Actual)
Dates: Start 2007-11; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
ACE/ARBs, ACE/ARBs+BB, hospitalisation rates, survival rate, reliability/ usability/applicability of computerised guideline, economic measurements | 2005 to 2007

CONTACTS AND LOCATIONS:
Overall Officials: Josep M Davins, MD, PhD, Principal Investigator — Unitat de Suport a la Recerca, Barcelona, Spain; Eva Frigola, Masters, Study Director — Unitat de Suport a la Recerca, Barcelona, Spain
Locations (1):
- Unitat de Suport a la Recerca, Barcelona, Spain